CLINICAL TRIAL: NCT03802916
Title: Safety and Acceptability of Deferiprone Delayed Release Tablets in Patients With Systemic Iron Overload
Acronym: TWICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Organization: Chiesi Canada Corp (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA61-0218
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Iron Overload Due to Repeated Red Blood Cell Transfusions
Keywords: iron overload; chelation; deferiprone; Ferriprox
MeSH Terms: conditions — Iron Overload | interventions — Deferiprone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dosage (Experimental): Patients in this group will receive a total daily dosage of deferiprone DR tablets that is closer to 75 mg/kg/day. The total dosage will be divided into two equal parts, taken about 12 hours apart.
  Interventions: Drug: Deferiprone DR tablets 1000 mg (Low dosage)
- High dosage (Experimental): Patients in this group will receive a total daily dosage of deferiprone DR tablets that is closer to 100 mg/kg/day. The total dosage will be divided into two equal parts, taken about 12 hours apart.
  Interventions: Drug: Deferiprone DR tablets 1000 mg (High dosage)

INTERVENTIONS:
Drug: Deferiprone DR tablets 1000 mg (Low dosage) — Deferiprone DR tablets 1000 mg
  Arms: Low dosage
Drug: Deferiprone DR tablets 1000 mg (High dosage) — Deferiprone DR tablets 1000 mg
  Arms: High dosage

SUMMARY:
Safety, tolerability, and acceptability of twice-daily dosing with deferiprone delayed-release (DR) tablets in patients with systemic iron overload.

DETAILED DESCRIPTION:
This study is looking at the safety, tolerability, and acceptability of twice-daily dosing with deferiprone delayed-release (DR) tablets in patients with systemic iron overload who are currently taking deferiprone immediate-release tablets (Ferriprox) three times a day. Ferriprox doses range from 75 milligrams per kilogram of body weight (mg/kg) per day to 100 mg/kg per day. Half the patients in the study will be on a dosage that is closer to the low end of the range, and half will be on a dosage that is closer to the high end. Both groups will be switched for one month to deferiprone DR tablets at approximately the same total daily dosage that they have been taking for Ferriprox.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years.
2. Diagnosis of thalassemia syndrome, sickle cell disease, or other disorder requiring a regular regimen of red blood cell transfusions.
3. On a stable regimen (≥3 months) of Ferriprox tablets for the treatment of systemic iron overload.
4. Absolute neutrophil count ≥1.5 x 10^9/L at screening.
5. A record of at least 12 measured alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels.

Exclusion Criteria:

1. Receipt of any iron chelator other than Ferriprox (i.e., combination therapy) in the last 3 months, or planning to receive it at any time during the period of the study.
2. ALT and/or AST value > 5 times the upper limit of normal (ULN) at screening
3. Active case of hepatitis B or C at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - New York Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
- St.Paul's Hospital, Vancouver, British Columbia, Canada
- National and Kapodistrian University of Athens, Aghia Sophia Children's Hospital, Goudi, Athens, Greece
- San Luigi Gonzaga University Hospital Reparto Microcitemie-Pediatria, Orbassano (TO), Regione Gonzole, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dosage | High Dosage
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient in the high-dosage group withdrew before receiving any study product
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dosage | High Dosage | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (9.9) | 40.4 (6.8) | 41.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Greece | 3 | 5 | 8
  Canada | 3 | 0 | 3
  United States | 1 | 2 | 3
  Italy | 8 | 7 | 16
Level of liver enzymes at baseline for low-dosage group [Mean (Standard Deviation); unit: units per liter] — Population: The results for this baseline measure are presented separately for each group.
  units per liter
    Baseline ALT: number analyzed (Participants) | 15 | 0 | 15
    Baseline ALT | 29.60 (19.88) |  | 29.60 (19.88)
    Baseline AST: number analyzed (Participants) | 15 | 0 | 15
    Baseline AST | 27.53 (10.00) |  | 27.53 (10.00)
Level of liver enzymes at baseline for high-dosage group [Mean (Standard Deviation); unit: units per liter] — Population: The results for this baseline measure are presented separately for each group.
  units per liter
    Baseline ALT: number analyzed (Participants) | 0 | 14 | 14
    Baseline ALT |  | 38.29 (22.43) | 38.29 (22.43)
    Baseline AST: number analyzed (Participants) | 0 | 14 | 14
    Baseline AST |  | 28.50 (11.39) | 28.50 (11.39)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients in Each Treatment Group Who Experience Post-dose Increases in Liver Enzyme Levels That Are Considered a Safety Concern.
Description: Levels of the liver enzymes alanine aminotransferase (ALT) and aspartate aminotransferase (AST) will be assessed throughout the study to determine if any patients have post-dose increases that are considered to be a safety concern. The criteria for being considered a safety concern are meeting one of the following:
  * For a patient whose level was within the normal range at baseline, the criterion is reaching a value of 5 times the upper limit of normal (ULN)
  * For a patient whose level was above the ULN at baseline, the criterion is reaching either 5 times the baseline value or 10 x ULN
Time Frame: Day 28
Population: One patient in the high-dosage group withdrew before providing any evaluable data
Measure: Count of Participants; unit: Participants
Groups:
- Low Dosage: Evaluable patients who received the lower dosage of deferiprone
- High Dosage: Evaluable patients who received the higher dosage of deferiprone
Arm/Group | Low Dosage | High Dosage
Number analyzed (Participants) | 15 | 14
Participants
  Patients with elevated ALT of clinical concern | 0 | 0
  Patients with elevated AST of clinical concern | 0 | 0

2. Secondary Outcome: The Percentage of Patients in Each Treatment Group Who Report Post-dose Occurrences of Gastrointestinal (GI) Distress.
Description: Patients will be asked to report any events of GI distress during the study, such as nausea, vomiting, diarrhea, abdominal pain, and dyspepsia.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dosage | High Dosage
Number analyzed (Participants) | 15 | 14
Participants | 3 | 3

3. Secondary Outcome: The Percentage of Patients in Each Group Who Indicate That They Prefer the Deferiprone DR Formulation Over the Immediate-release Formulation.
Description: At the end of the study, patients will complete a questionnaire to indicate which formulation they prefer.
Time Frame: Day 28
Population: One of the evaluable patients withdrew before completing the questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Low Dosage; High Dosage: Patients who completed the questionnaire
Arm/Group | Low Dosage | High Dosage
Number analyzed (Participants) | 15 | 13
Participants | 13 | 13
Statistical Analysis 1: Comparison: Low Dosage; One-sample proportion test to determine if the overall preference for deferiprone DR was greater than chance (i.e., a 50% preference for each formulation); Test type: Superiority; p = 0.0074, One-sample proportion test — A p-value was calculated for the one-sample proportion test
Statistical Analysis 2: Comparison: High Dosage; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0002, One-sample proportion test — A p-value was calculated for the one-sample proportion test

ADVERSE EVENTS:
Time Frame: Baseline to Day 28
Arm/Group | Low Dosage | High Dosage
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 10/15 | 9/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dosage (N=15) | High Dosage (N=14)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (5)
Migraine (Nervous system disorders) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03802916/Prot_SAP_002.pdf